CLINICAL TRIAL: NCT02437708
Title: Regenerative Endodontic Procedure of Immature Permanent Teeth With the Use of Autologous L-PRF: a Pilot Controlled, Clinical Trial
Brief Title: Regenerative Endodontic Procedure of Immature Permanent Teeth With L-PRF: a Pilot Controlled, Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S56810 (ML10723) B322201421941
Record Dates: First submitted 2015-05-04; First posted 2015-05-08 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Endodontic Inflammation
Keywords: regenerative endodontics; platelet rich fibrin
MeSH Terms: conditions — Pulpitis | interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- REP with L-PRF (Experimental): The first REP session will be performed as described by Diogenes et al. (2013). For the second REP-session a venipunction will be performed before the endodontic treatment. 2 to 4 tubes of blood will be collected per tooth. These blood samples will be put into a centrifuge for 12 minutes at 2700 rpm. Fibrin clots will be collected after centrifugation and inserted in the root canal with endodontic pluggers. Medcem Portlandcement (GmbH, Swiss) will be used instead of mineral trioxide aggregate in the second session, to prevent tooth discoloration.
  Interventions: Procedure: REP with L-PRF; Biological: stem and progenitor cells
- REP (Active Comparator): A REP will be performed on immature infected permanent teeth, as described in the protocol of Diogenes et al. (2013). Medcem Portlandcement (GmbH, Swiss) will be used instead of mineral trioxide aggregate in the second session, to prevent tooth discoloration.
  Interventions: Procedure: REP

INTERVENTIONS:
Procedure: REP with L-PRF
  Arms: REP with L-PRF
Procedure: REP
  Arms: REP
Biological: stem and progenitor cells
  Arms: REP with L-PRF

SUMMARY:
This study evaluates the impact of autologous 'leucocyte and platelet rich fibrin' (L-PRF) on the periapical bone healing and further root development of infected immature permanent teeth. In the test group regenerative endodontic procedure (REP) is performed with L-PRF as scaffold, in the control group REP without L-PRF is performed .

DETAILED DESCRIPTION:
Regenerative endodontic procedures are biologically based procedures designed to restore function of a damaged and nonfunctioning pulp by stimulation of existing stem and progenitor cells present in the root canal and/or the introduction and stimulation of new stem and dental pulp progenitor cells into the root canal under conditions that are favorable to their differentiation and reestablishment of function. L-PRF has the potential advantage of creating a bioactive construct that stimulates the local environment for differentiation and proliferation of these stem and progenitor cells. We have designed this confirmatory study to test the hypothesis that the use of L-PRF in REP of infected permanent immature teeth will accelerate periapical bone healing and stimulate the root maturation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed Consent
* Permanent immature teeth with weak root canal walls (hopeless prognosis)
* Patients younger than 25 years

Exclusion Criteria:

* - Unlikely to be able to comply with the study procedures, as judged by the investigator.
* Patients older than 25 years
* Deciduous teeth
* Permanent (immature) teeth that can be treated by a "regular" root canal treatment/ apexification
* Known or suspected current malignancy
* History of chemotherapy within 5 years prior to study
* History of radiation in the head and neck region
* History of other metabolic bone diseases
* A medical history that makes REP unfavorable
* Involvement in the planning and conduct of the study
* Previous enrolment in the present study

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2014-09; Primary Completion 2019-08 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Amount of periapical bone healing, measured on intra-oral bidimensional radiographs. | 3 years

SECONDARY OUTCOMES:
Amount of root development or maturogenesis,by measuring: | 3 years
  on intra-oral bidimensional radiographs: the increase in root canal wall thickness.
Amount of root development or maturogenesis,by measuring: | 3 years
  on intra-oral bidimensional radiographs: the increase in root canal length.

OTHER OUTCOMES:
On conebeam CT (tridimensional measuring): the amount of periapical bone healing, increase in root canal wall thickness and root canal length. (composite) | 3 years
Patient related outcome, measured by a questionnaire | 3 years
Patient related outcome, measured by a pain-scale | 3 years
Microbial diversity in the infected immature root canal | intraoperative
  Q-PCR analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lambrechts, Prof, Dr, Principal Investigator — Department of Oral Health Sciences, KU Leuven & Dentistry, University Hospitals Leuven, Belgium
Locations (4):
- Belgium (4):
  - Megabite Dental Office, Brussels
  - C-Endo, Herent
  - Department of Oral Health Sciences, KU Leuven & Dentistry, University Hospitals Leuven, Leuven
  - EndoVanGorp, Rotselaar

REFERENCES:
- [Background] Diogenes A, Michael AH, Teixeira FB, Hargreaves KM. An update on clinical regenerative endodontics. Endod Top. 2013;28:2-23.